CLINICAL TRIAL: NCT00333008
Title: Phase II Dose Study of Doxil in a Dose Dense, 14 Day CDOP/Rituximab Regimen for Patients With Diffuse Large B-Cell NHL > 60 Years or With Compromised Cardiac Status
Brief Title: A Dose Study of Doxil in a Dose Dense, 14 Day CDOP/Rituximab Regimen for Patients With Diffuse Large B-Cell Non-Hodgkin Lymphoma (NHL)> 60 Years or With Compromised Cardiac Status.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Alvin and Lois Lapidus Cancer Institute (Other)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY-012006
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2006-09-26 (Estimated); Status verified 2006-09

CONDITIONS: Diffuse Large B Cell Lymphoma; Lymphoma, Non-Hodgkin
Keywords: Diffuse Large B Cell Lymphoma; CDOP; Dose Dense; Anne Arbor Stage I-IV; Any IPI score
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — liposomal doxorubicin; Cyclophosphamide; Vincristine; Prednisone; Rituximab; pegfilgrastim

INTERVENTIONS:
Drug: Doxil
Drug: Cyclophosphamide
Drug: Vincristine
Drug: Prednisone
Drug: Rituximab
Drug: Pegfilgrastim

SUMMARY:
The purpose of this study is to evaluate the feasibility and tolerability of delivering a full dose, on time schedule of dose-dense CDOP-R (cyclophosphamide, doxil, vincristine, prednisone, and rituximab) in NHL.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most frequent type of non-Hodgkin's lymphoma with more than half of the patients being over the age of 60 years. Elderly patients with cancer are defined by the American Society of Clinical Oncology as a "special population" due to their disease characteristics, additional health problems, and need for aggressive supportive care strategies to reduce morbidity and mortality. The combination of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) remains as standard therapy for the treatment of DLBCL, but elderly patients tend to tolerate the CHOP therapy less when compared to younger patients. Cardiac toxicity, as well as decrease in blood counts, are the most common side effects in the elderly population. For these reasons, many doctors are reluctant to use standard combinations and doses of chemotherapy in the elderly for fear of increased morbidity. DLBCL in the elderly is also somewhat unique in that the elderly patients appear to have more aggressive disease and poor overall outcome. In order to maximize the tolerability of treatment and thus potentially enhance overall treatment success in this population, it is necessary to look at alternative treatments. This clinical trial is based on currently accepted standard NHL therapy (CHOP-Rituximab) in which Doxil is substituted for Adriamycin. Growth factor will be used for support of acceptable blood counts. Chemotherapy regimens that include rituximab are now the gold standard for treatment of DLBCL. If indeed, delivering full dose chemotherapy without treatment delays leads to higher remission and cure rates, then this offers a significant proportion of NHL patients who are elderly a chance for cure rather than providing treatment for comfort measures while preserving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old and older or 18 years old and older with significant/potential cardiac morbidity
* Diagnosis of diffuse large B cell lymphoma, Ann Arbor stage I-IV, any International Prognostic Index (IPI) score.
* Previously untreated
* New York Heart Association (NYHA) classification of Class III or better
* Baseline ejection fraction (EF) > 25%
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3
* Unless attributable to NHL: absolute neutrophil count (ANC) > 1500/uL, platelets > 100,000/uL; hemoglobin > 9.0 g/dl
* Bilirubin < 1.5 mg/dL (unless related to lymphoma)
* Hepatic: transaminases < 2.5 x upper limit of normal (ULN) (unless related to lymphoma)
* Creatinine < 2.5 mg/dl (unless related to lymphoma)

Exclusion Criteria:

* No HIV+ individuals
* No primary central nervous system (CNS) lymphoma
* No pregnant or lactating women
* No serious active infection
* History of prior malignancy within the last 5 years other than subject's original cancer diagnosis listed in inclusion criteria with the exception of curatively treated basal cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2006-05

PRIMARY OUTCOMES:
Safety assessment: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTACAE) v3.0
Efficacy: tumor evaluations every three (q 3) cycles

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Noga, MD, PhD, Principal Investigator — Sinai Hospital of Baltimore, The Alvin and Lois Lapidus Cancer Institute
Locations (2):
- United States (2):
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland